CLINICAL TRIAL: NCT06037278
Title: MyPAO Patient Specific Guides and Surgical Planning for Periacetabular Osteotomy; Post Marketing Evaluation Study
Brief Title: Patient Specific Guides and Surgical Planning for Periacetabular Osteotomy; Post Marketing Evaluation Study
Acronym: MyPAO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Royal Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROH22ORTH13
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Pelvic Osteotomy; Acetabular Dysplasia; Periacetabular Osteotomy
Keywords: Customised surgical guides
MeSH Terms: conditions — Hip Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MyPAO use (Other): SIngle arm study, use of device
  Interventions: Device: MyPAO

INTERVENTIONS:
Device: MyPAO — use of MyPAO surgical guide to support periacetabular osteotomy procedures for treatment of acetabular dysplasia
  Other Names: periacetabular osteotomy

SUMMARY:
A case series to provide post marketing evaluation of the MyPAO surgical planning and patient specific guides technology. This will be a single-centre, multi-surgeon evaluation assessing the safety of the use of these guides in periacetabular osteotomy surgery.

DETAILED DESCRIPTION:
After enrolment, baseline data will be collected including age, sex and ethnicity of the participant. The radiographic measures of centre edge angle of Wiberg and acetabular inclination will be measured by the surgeon and patient reported outcome measures (PROMS) will be collected. The PROMS collected at usual care timepoints in patients undergoing pelvic osteotomy will be collated for use in the dataset. Peri-operative data, including clinician opinion on ease of use, intraoperative dose of radiation used and device associated adverse events, will be recorded and reported in the results.

ELIGIBILITY:
Inclusion Criteria:

* · Age greater than 18 years

  * Patient undergoing pelvic osteotomy

Exclusion Criteria:

* · Evidence of hip degeneration assessed by the surgeon on x-ray (Tonnis Grade 1 or greater)

  * Known allergy to Polyamide PA12
  * Unable to provide written informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Product safety assessment | 3 months post-surgery
  evaluate the use of the MyPAOTM technology by reviewing number of device related adverse events, in order to continue to assess product safety as part of post marketing surveillance.

SECONDARY OUTCOMES:
Proof of concept | 12 months
  surgeon questionnaires after each case. We will determine technical difficulties in using the device, surgeon satisfaction with the use of guides and the guided correction and the presence of any intra-operative adverse events.
i-hot12 questionnaire | 12 months post-surgery
  hip-specific health related quality of life outcome tool
Eq-5D | 12 months post-surgery
  validated measure of health-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Orthopaedic Hospital NHS Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No